CLINICAL TRIAL: NCT05490589
Title: Evaluation of the Implementation of a Parenting Program in Parents With Children Aged 4 to 12 Years and One Parent With an Alcohol Use Disorders
Acronym: APPROCHILD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC20.0173
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Addiction, Alcohol
Keywords: Alcohol dependance
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EQUIPE Program (Experimental)
  Interventions: Other: EQUIPE Program

INTERVENTIONS:
Other: EQUIPE Program — EQUIPE is a manualised group community-based parent education programme. Groups consist of 15 parents who meet with one or two trained group leaders for weekly 2-hour sessions over 10 weeks.
  This program promotes skill development in parents, strengthens relationships with children, increases cooperation, and helps solve problems in the home.

SUMMARY:
Alcohol use disorders are a major public health problem in Europe. The average prevalence of Alcohol Use Disorders (AUD) in the general population is 7.5%, although there are large variations between countries. According to the literature, 20 to 30% of children have parents with problematic alcohol use. Public health authorities are alarmed by the precociousness of alcohol consumption in the youngest age and by the prevalence of alcohol consumption in adolescence. One of the well-established risk factors for alcohol use and abuse is having a parent with AUD. Compared with people growing up without any parent with AUD, the relative risk of suffering negative life events in childhood is 2 to 13 times higher if one or both parents have alcohol use disorders. A family history of Alcohol Use Disorders is predictive of earlier alcohol, tobacco, or cannabis use in adolescence, but it is also associated with a higher risk of developing substance use disorders.

DETAILED DESCRIPTION:
Despite these alarming data, very few studies have focused on preventing alcohol use in vulnerable populations with at least one parent with Alcohol Use Disorders. Parenting support programs have been developed, according to current knowledges, there are no programs in French that target families with Alcohol Use Disorders.

The EQUIPE program is a French adaptation of the Canadian program, Community Parent Education (COPE). It is a psycho-educational intervention program developed́ by C. Cunningham (McMaster University, Hamilton, ON). It is aimed at improving parenting skills. Its format involves a 2 hr/week session and is spread over 10 weeks. During the sessions, using short video vignettes, parents are encouraged to find their own solutions to difficulties in managing their child's behaviour. These solutions are then discussed among parents in the presence of professionals (animators or facilitators). Finally, educational strategies are adopted and practiced in the family setting. This program aims to strengthen the protective factors of children in the face of risky behaviours that they may develop during adolescence, by having parents and children work together on communication, the establishment of warm and positive relationships and their ability to resolve problems and conflicts. This EQUIPE program has been evaluated in Quebec with families experiencing difficulties with children with behavioral problems. At present, in France, no parenting support program is applied to families with addictive behaviors in a broad and evaluated manner. The investigators believe that an "early" intervention could allow to apprehend future social and mental problems (malaise and depression, school dropout, delinquency...), and limit the risks of intra-family conflicts and thus reduce the negative impact on the potential development of psychological disorders and addictive behaviors in adolescence and adulthood. The implementation of this parenting support program, applied to families suffering from alcohol addictive behaviors and at an early stage with children aged 3-12 years, would seem to be relevant in order to reinforce parenting skills.

ELIGIBILITY:
Inclusion Criteria :

* Major subject (age > 18 years)
* Patient with a child between 4 and 12 years old
* Patient living with his/her child permanently or partially
* Patient or his/ her spouse with an alcohol use disorder (at least 3 of the 11 DSM 5 criteria for alcohol use disorder in the past 12 months)
* Written and informed consent

Exclusion Criteria :

* Minor subject (age < 18 years)
* Acute, unstabilized psychiatric disorder impairing judgment
* Incapacity or refusal to give consent
* Subject under judicial protection or family habilitation
* Subject deprived of liberty by judicial or administrative decision, under guardianship or curatorship ;
* Non comprehension of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2027-08-22 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a parenting program | At 6 month post EQUIPE program
  Overall score measuring the level of parental stress, obtained using the Parental Stress Index (PSI), measured at the post-inclusion visit and at the 6-month post-program visit.
  Parental Stress Index was designed to evaluate the magnitude of stress in the parent-child system, with 101-item inventory that focuses on two major domains of stress: child characteristics and parent characteristics.
  The score is obtained by summing the responses to the items and then converting it to a percentile. A high score means that the parent is stressed.

SECONDARY OUTCOMES:
Score on the different domains of the Parental Stress Index | At 6 month post EQUIPE program
  The different domains of the Parental Stress Index were :
  * Within the Child Domain, six subscales (Distractibility/Hyperactivity, Adaptability, Demandingness, Reinforces Parent, Acceptability and Mood)
  * Within the Parent Domain, seven subscales (Competence, Isolation, Attachment, Health, Role Restriction, Depression, and Spouse/Parenting Partner Relationship)
  * The Total Stress scale is combined of the two domains (Child and Parent).
Evaluation of self-esteem | At 3, 6 and 12 month post EQUIPE program
  Self-esteem is evaluated by the Rosenberg scale. The Rosenberg Self-Esteem Scale measures overall self-confidence by measuring both positive and negative feelings. The scale has 10 items. Each item is measured on a scale of 1 to 4, from strongly disagree for 1 to strongly agree for 4.
Evaluation on children's behaviors | At 3, 6 and 12 month post EQUIPE program
  For assessed the impact on children's behaviors, Strengths and Difficulties Questionnaire (SDQ) was used. SDQ is a questionaire which used for mental health problems screening in children. This questionnaire measures the presence of behaviours that indicate emotional difficulties such as physical aggression, isolation, anxiety, difficulty concentrating and impulsivity. It is intended for children from 3 to 16 years old and can be completed by the parent. SDQ includes 25 questions that the parent can answer with "not true", "somewhat true" or "very true". The score is obtained as follows: for each statement, the answer "false" gives zero points, "somewhat true" one point and "absolutely true" two points. With the exception of the items marked in bold, for which the "false" answer gives two points and the "absolutely true" answer zero, the other option remains the same. Emotional or behavioral difficulties are considered to exist when the score is 16 or higher.
Evaluation of alcohol use | At 3, 6 and 12 month post EQUIPE program
  Alcohol consumption measured by the Alcohol Timeline Followback (ATLFB) score at each visit. The A-TLFB is a method of assessing alcohol consumption that provides an estimate of the daily amount of alcohol consumed in standard units.It has been evaluated in clinical and non-clinical populations and in adults and adolescents. It is in the form of a calendar. Respondents report their daily alcohol consumption over a specified period of the past 30 days. Recall aids can be used during the completion of the questionnaire (dates, events, etc.). This tool has good psychometric qualities and is recommended when precise information on the quantities of alcohol consumed or the number of days of consumption is needed.
  It allows to identify the number of days of alcohol consumption in the month and the number of days with alcohol consumption above 5 standard units/d.
  No score is obtained but we have the follow-up of the patients' consumption
Evaluation of severity of alcohol use disorders | At 3, 6 and 12 month post EQUIPE program
  Severity of alcohol use disorders at each visit, as measured by the number of Diagnostic and Statistical manual of Mental disorders 5 (DSM5) criteria. The DSM5 score is diagnosis of addiction is based on well-defined criteria set out in the Diagnostic and Statistical manual of Mental disorders (DSM), the fifth edition of which was published in 2013. The questionnaire consists of 11 items (diagnostic criteria for substance use disorders from the American Psychiatric Association's DSM V). The presence of 2 to 3 criteria: low addiction / Presence of 4 to 5 criteria: moderate addiction / Presence of 6 or more criteria: severe addiction.
Evaluation of the progression of anxiety and depressive symptoms | At 3, 6 and 12 month post EQUIPE program
  Evaluation of the progression of anxiety and depressive symptoms This evolution will be assessed by Hopkins Symptom Checklist (HSCL25). The HSCL-25 is a questionnaire, consisting of 25 questions relating to the presence and intensity of symptoms of anxiety (question ranging from 1 to 10) and depression (question ranging from 11 to 25) during the last full week. The patient is asked to rate each item on a four-point scale, ranging from 1: strongly disagree, to 4: strongly agree. To obtain the diagnostic score, the responses to all questions are summed and divided by 25.
Evaluation of the quality of life during the follow-up time | At 3, 6 and 12 month post EQUIPE program
  Quality of life evaluated by the World Health Organization Quality of Life (WHOQOL scale brief). The WHOQOL-BREF instrument consists of 26 items that measure the following broad domains: physical health, psychological health, social relationships and environment. It is used to assess the quality of life of adults.
  Each question is scored on a 5-point Likert scale (1 to 5). The sum of the points gives us the score. The higher the score, the better the patient's quality of life
Evaluation of acceptability of the study by the participants | At 3 month post EQUIPE program
  Acceptability will be assessed using a Likert scale that asks individuals about their level of agreement or disagreement with a statement. The question "Do you think your participation in the EQUIPE program was useful to you?" will be asked at the end of the program.
  Free comments will be left open with a question "Do you have any comments on the program?"

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 42 month and ending 15 years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of BrestUH. Requestors will be required to sign and complete a data access agreement.